CLINICAL TRIAL: NCT01652976
Title: Phase II Study of 5-Fluorouracil, Oxaliplatin Plus Dasatinib (FOLFOX-D) in First-line Metastatic Pancreatic Adenocarcinoma
Brief Title: Phase II Study of 5-FU, Oxaliplatin Plus Dasatinib in Metastatic Pancreatic Adenocarcinoma
Acronym: FOLFOX-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600540; CA180-359 (Other: University of Florida); OCR11303 (Other: OnCore)
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: Metastatic; Pancreatic Cancer; Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms; Adenocarcinoma | interventions — Dasatinib; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Dasatinib and mFOLFOX6
  Interventions: Drug: Dasatinib; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 150mg PO daily on days 1-14 of each 14 day cycle
  Other Names: Sprycel
Drug: mFOLFOX6 — mFOLFOX6 (oxaliplatin 85mg/m2 IV, leucovorin 400mg/m2 IV, 5-Fluorouracil bolus 400mg/m2 IV, and 5-Fluorouracil 2400mg/m2 IV) on day 1 of each 14 day cycle
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil

SUMMARY:
The purpose of this research study is to determine if the study drug, dasatinib, given in combination with 5-Fluorouracil, leucovorin and oxaliplatin (FOLFOX) will work against metastatic pancreatic cancer.

Dasatinib is a Food and Drug Administration (FDA) approved drug for treating chronic myelogenous leukemia and acute lymphoblastic leukemia, however it is not currently approved for use in the treatment of pancreatic cancer.

DETAILED DESCRIPTION:
Systemic control of pancreatic cancer remains a clinical unmet need. The recent superiority of 5-FU based combination therapies over the historical standard gemcitabine represents an opportunity to develop novel combinations of synergistic and effective cytotoxic and biologic targeted therapies. Src excess activity has been demonstrated in pancreatic cancer and is implicated in the invasive and metastatic phenotype clearly represented by this disease. Inhibition of Src activity is associated with numerous biologic modifications capable of positively modifying this phenotype and appears to have synergy with restoring inherent chemosensitivity. The addition of dasatinib to FOLFOX (FOLFOX-D) represents a novel therapeutic regimen in pancreatic cancer with safety and pharmacokinetic data already having been established in colorectal cancer. This protocol will test the safety and activity of this combination in pancreatic cancer where current clinical outcomes remain far from optimal.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic adenocarcinoma with evidence of metastatic disease on imaging
* Measurable disease (per RECIST 1.1)
* ECOG Performance Status 0-2
* No prior chemotherapy or radiotherapy for metastatic pancreatic cancer. Patients may have received prior treatment for non-metastatic disease; however the diagnosis of metastatic disease must have been made more than 6 months after completion of treatment.
* Patients may have a history of other malignancies if there is no current evidence of persistent or recurrent disease and they are not undergoing any active therapy (including hormonal)
* Patent biliary system
* Patients receiving anti-coagulation treatment with an agent such as Coumadin or heparin may be allowed to participate, provided they are on stable anti-coagulation therapy with no active bleeding and have no condition that carries a high risk of bleeding
* Adequate organ and marrow function
* Ability to take oral medication (dasatinib must be swallowed whole)
* Patient agrees to discontinue prohibited concomitant medications
* Age > 18 years
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception throughout the study and for at least 4 weeks after the last dose of study drug.
* A male subject of fathering potential must use an adequate method of contraception throughout the study and for at least 4 weeks after the last dose of study drug.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after the last dose of study drug. Women who are pregnant or breastfeeding and sexually active fertile men not using effective birth control if their partners are WOCBP are also excluded.
* History of known brain metastases or carcinomatous meningitis
* Recent major surgery (within 4 weeks) or minor surgery (within 2 weeks), excluding placement of a vascular access device or biliary stent
* Uncontrolled diabetes
* Any sensory neuropathy > grade 1 at baseline
* Serious active or uncontrolled infection
* Concurrent medical condition which may increase the risk of toxicity including clinically significant pleural or pericardial effusion, patients with known DPD deficiency or patients with a history of allergic reactions attributed to oxaliplatin, 5-FU or leucovorin.
* Cardiac Symptoms including unstable angina or stable angina markedly limiting ordinary physical activity, NYHA class III or IV congestive heart failure, myocardial infarction or stroke within 6 months of study enrollment, diagnosed congenital long QT syndrome, any history of clinically significant ventricular arrhythmias, prolonged QTc interval on pre-entry ECG or clinically significant peripheral vascular disease.
* Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
* History of significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders, diagnosed acquired bleeding disorder within one year or ongoing or recent (≤ 3 months) significant gastrointestinal bleeding.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy, might affect the interpretation of the results of the study, or that puts the subject at high risk for treatment complications.
* Use of category I drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Use of potent CYP3A4 inhibitors that significantly increase dasatinib exposure
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J George, Jr., MD, FACP, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] George TJ Jr, Trevino JG, Liu C. Src inhibition is still a relevant target in pancreatic cancer. Oncologist. 2014 Feb;19(2):211. doi: 10.1634/theoncologist.2013-0410. Epub 2014 Jan 23. No abstract available. PMID 24457377

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib and mFOLFOX6: Dasatinib and mFOLFOX6
  Dasatinib: Dasatinib 150mg PO daily on days 1-14 of each 14 day cycle
  mFOLFOX6: mFOLFOX6 (oxaliplatin 85mg/m2 IV, leucovorin 400mg/m2 IV, 5-Fluorouracil bolus 400mg/m2 IV, and 5-Fluorouracil 2400mg/m2 IV) on day 1 of each 14 day cycle
Period: Overall Study
Arm/Group | Dasatinib and mFOLFOX6
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 65 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44
ECOG Performance status [Count of Participants; unit: Participants] — ECOG performance status describes a patient's level of functioning in terms of daily activity level and how capable they are of self-care on a scale of 0 (best)-5 (worst). The meaning of each performance status grade reported at baseline is below:
  0 = Normal activity
  1. = Fully active, able to carry on all pre-disease performance without restriction; Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature
  2. = In bed < 50% of the time; ambulatory and capable of all self-care, but unable to carry out any work activities
  Participants
    Status = 0 | 22
    Status = 1 | 19
    Status = 2 | 2
    Performance Status Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Determine activity of 5-Fluorouracil, leucovorin, and oxaliplatin (FOLFOX) plus dasatinib on progression free survival (PFS) in patients with metastatic pancreatic adenocarcinoma
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
months | 4 [2.3 to 8.5]

2. Secondary Outcome: Response Rate
Description: To determine the response rate (RR) by RECIST 1.1 criteria. The response rate is the number of subjects who had either a complete or partial response by RECIST 1.1 criteria. RECIST 1.1 criteria defines a partial response as a decrease of the sum of the largest diameter each target lesion by at least 30%. A complete response is defined as the disappearance of all target lesions (except lymph nodes, whose short axis must measure 10 mm or less). The imaging modality used for all RECIST assessments in this study was CT.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
percentage of subjects | 25 [13.19 to 40.34]

3. Secondary Outcome: Freedom From Metastasis
Description: To determine the rate of freedom from metastasis (FFM), which is defined as the percentage of subjects with documented progressive disease (by RECIST 1.1 criteria) who had no new lesions. RECIST 1.1 criteria defines progressive disease as the appearance of one or more new lesions and/or the increase of the sum of the largest diameter of the target lesions by at least 20% from the smallest sum collected (the sum must also have increased by at least 5 mm).
Time Frame: 3 years
Population: The number of participants analyzed for this outcome measure only includes the 29 participants who had documented disease progression (by RECIST 1.1 criteria) during study participation.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 29
percentage of subjects | 65.5 [45.7 to 82.1]

4. Secondary Outcome: Median Time To Progression
Description: To determine the median time to progression (TTP). TTP is defined as the time (in months) from when a subject achieves either a complete or partial response by RECIST 1.1 criteria until progressive disease (by RECIST 1.1 criteria) or death occurs.
Time Frame: 3 years
Population: The number of participants analyzed for this outcome measure includes only the 11 participants who achieved either a complete or partial response by RECIST 1.1 criteria during study participation.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 11
months | 9.8 [8.6 to 19.5]

5. Secondary Outcome: Median Overall Survival
Description: To determine median overall survival (OS) in months
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
months | 10.6 [6.9 to 12.7]

6. Secondary Outcome: Clinical Benefit Rate
Description: To determine the clinical benefit rate (CBR). The CBR is defined as the percentage of subjects who achieved either a complete or partial response or stable disease by RECIST 1.1 criteria. RECIST 1.1 criteria defines a partial response as a decrease of the sum of the largest diameter each target lesion by at least 30%. A complete response is defined as the disappearance of all target lesions (except lymph nodes, whose short axis must measure 10 mm or less). By RECIST 1.1 criteria, a subject is considered to have stable disease when the sum of the largest diameter of the target lesions has neither decreased enough to qualify as a partial response not increased enough to qualify as progressive disease.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
percentage of subjects | 56.82 [41.03 to 71.65]

7. Secondary Outcome: Site of Failure
Description: To determine the site of failure of this regimen in this population. The site of failure is the anatomical site(s) where disease progression by RECIST 1.1 criteria was noted on imaging.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
Participants
  Left pleural effusion | 1
  Liver | 12
  Lungs | 3
  Pancreas/liver | 4
  Peritoneal carcinomatosis | 1
  peritoneal carcinomatosis/liver | 1
  Spleen/liver | 1

8. Secondary Outcome: Safety and Tolerability
Description: To determine the safety profile and tolerability of this regimen in this population by evaluating acute treatment related toxicities using CTCAE v4.0 criteria. Using the CTCAE v4.0, the severity of each adverse event reported was graded on a scale of 1 (mild severity) to 5 (fatal). For this outcome measure the percentage of subjects experiencing any adverse event of each CTCAE grade was tabulated.
Time Frame: 3 years
Measure: Number; unit: percentage of subjects
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
percentage of subjects
  Percent of subjects experiencing a Grade 1 event | 88.6
  Percent of subjects experiencing a grade 2 event | 90.9
  Percent of subjects experiencing a Grade 3 event | 86.4
  Percent of subjects experiencing a Grade 4 event | 22.7
  Percent of subjects experiencing a grade 5 event | 9.1

9. Secondary Outcome: Drug Compliance
Description: To determine patient compliance with oral therapy. For this outcome measure, compliance with oral therapy is defined as the percentage of subjects that took dasatinib for at least one cycle. Compliance with oral therapy was documented with a medication diary that subjects were asked to complete to document whether each dose of dasatinib was taken.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
percentage of subjects | 93.2 [81.3 to 98.6]

10. Secondary Outcome: Quality of Life, as Measured by the Cancer Therapy Satisfaction Questionnaire (CTSQ), 2007
Description: To determine the quality of life (QOL) of patients receiving this therapy using the CTSQ questionnaire. The CTSQ consists of 16 questions where subjects respond with a score on a scale of 0 (worst)-4 (best). The responses to the questions are used to calculate 3 subscores: Expectations of Therapy (ET), Feelings about Side Effects (FSE), and Satisfaction with Therapy (SWT). Each subscore is calculated by multiplying the mean response value for the questions used to calculate that subscore by 25. The maximum value is 100 and the minimum value is 0 for all 3 subscores. A higher subscore indicates better QOL in that area. The mean difference in each of the 3 subscores from baseline and 95% confidence interval for the entire study population is reported here. A negative mean difference indicates a decrease from baseline in QOL for that area.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
score on a scale
  Subscore difference for ET | -8.4 [-16.5 to -0.4]
  Subscore difference for FSE | 2.1 [-8.1 to 12.3]
  Subscore difference for SWT | -0.5 [-8.8 to 7.8]

11. Secondary Outcome: Quality of Life, as Measured by the Functional Assessment of Chronic Illness Therapy; Hepatobiliary Cancer (FACT-Hep) Questionnaire (Version 4.0)
Description: The FACT-Hep consists of 45 questions where subjects respond with a score on a scale of 0 (worst)-4 (best). The responses to the questions are summed to calculate 5 subscores: Physical Well-Being (PWB), Social Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB), and Hepatobiliary Cancer Subscale (HCS). The mean difference in each of the 5 subscores from baseline, as well as the total score of the 5 subscores (the FACT-Hep Total Score) for the entire study population is reported here. The mean difference in the FACT-G Total Score (calculated by summing the PWB, SWB, EWB, and FWB subscores) is also reported here. A negative mean difference indicates a decrease from baseline in QOL. Score ranges- PWB subscore: 0-28, SWB subscore: 0-28, EWB subscore: 0-24, FWB subscore: 0-28, HCS subscore: 0-72, FACT-G Total Score: 0-108, and FACT-Hep Total Score: 0-180. A higher value for each subscore or total score indicates better QOL.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dasatinib and mFOLFOX6
Number analyzed (Participants) | 44
score on a scale
  Subscore difference for PWB | -4.4 [-6.7 to -2.1]
  Subscore difference for SWB | -0.9 [-2.5 to 0.8]
  Subscore difference for EWB | 0.6 [-1.1 to 2.3]
  Subscore difference for FWB | -2.8 [-4.6 to -1.0]
  Subscore difference for HCS | -6.3 [-9.3 to -3.4]
  Difference in FACT-G Total Score | -7.4 [-11.9 to -2.9]
  Difference in FACT-Hep Total Score | -13.7 [-20.0 to -7.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time that informed consent was signed until 30 days after the last dose of study treatment. During this time frame, adverse event data was collected at the time informed consent was signed, on day 1 of each treatment cycle, and 30 days after the last dose of study treatment at a minimum. The time over which adverse event data was collected for the subjects ranged from 8 days to 44 months, an average of 8.5 months.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator at the time informed consent was signed, on day 1 of each treatment cycle, and 30 days after the last dose of study treatment at a minimum. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 42/44
Serious Adverse Events (participants affected / at risk) | 24/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=44)
Nervous system disorders, other (Stroke-like symptoms) (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Gastrointestinal disorders, other (gastrointestinal hemorrhage-unknown site) (Gastrointestinal disorders) | 1
Abdominal infection (Gastrointestinal disorders) | 1
Renal and urinary disorders, other (kidney stone) (Renal and urinary disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Fever (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Acute renal injury (Renal and urinary disorders) | 1
Flu-like symptoms (General disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subdural hematoma (Nervous system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Cholangitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Respiratory, thoracic, and mediastinal disorders, other (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal infection (Gastrointestinal disorders) | 1
Oral Mucositis (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Wound dehiscense (Injury, poisoning and procedural complications) | 1
Edema trunk (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=44)
Vomiting (Gastrointestinal disorders) | 26
Urinary frequency (Renal and urinary disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Skin and subcutaneous disorders, other (Skin and subcutaneous tissue disorders) | 5
Weight Loss (Investigations) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Platelet count decreased (Investigations) | 8
Peripheral sensory Neuropathy (Nervous system disorders) | 30
Periorbital edema (Skin and subcutaneous tissue disorders) | 6
Parasthesia (Nervous system disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 3
Oral Pain (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 15
Nausea (Gastrointestinal disorders) | 31
Mucositis oral (Gastrointestinal disorders) | 17
Localized edema (General disorders) | 3
Insomnia (Psychiatric disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hemorrhoids (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 6
General disorders and administrative site conditions - other (General disorders) | 3 — Night sweats
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Flu-like symtoms (General disorders) | 4
Fever (General disorders) | 11
Fatigue (General disorders) | 32
Fall (Injury, poisoning and procedural complications) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Edema limbs (General disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Dysgeusia (Nervous system disorders) | 12
Dysethesia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 7
Diarrhea (Gastrointestinal disorders) | 24
Depression (Psychiatric disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Constipation (Gastrointestinal disorders) | 19
Chills (General disorders) | 5
Bloating (Gastrointestinal disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Ascites (Gastrointestinal disorders) | 5
Anxiety (Psychiatric disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 21
Anemia (Blood and lymphatic system disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT01652976/Prot_SAP_000.pdf